CLINICAL TRIAL: NCT07402850
Title: Oscillating Positive Expiratory Pressure Therapy Versus Autogenic Drainage in Patients With Chronic Obstructive Pulmonary Disease: Effects on Pulmonary Function, Sputum Clearance, Dyspnea, and Quality of Life
Brief Title: Oscillating Positive Expiratory Pressure Therapy Versus Autogenic Drainage in Patients With COPD
Acronym: OPEP-AD-COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adnan Hashim (Other)
Responsible Party: Sponsor-Investigator, Adnan Hashim, Doctor of Physical Therapy Student, University of Lahore
Organization: University of Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHRI/IREB/26/01/0079
Record Dates: First submitted 2026-01-26; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Airway Clearance
Keywords: COPD; Oscillating Positive Expiratory Pressure; Autogenic Drainage; Physiotherapy; Pulmonary Rehabilitation; Airway Clearance Techniques
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Participants were allocated into two parallel groups to receive either oscillating positive expiratory pressure therapy or autogenic drainage for a four-week intervention period.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blinded to group allocation to minimize assessment bias. Participants and care providers were not blinded due to the nature of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oscillating Positive Expiratory Pressure Therapy Group (Experimental): Participants in this group received oscillating positive expiratory pressure therapy as an airway clearance technique for four weeks.
  Interventions: Device: Oscillating Positive Expiratory Pressure Therapy
- Autogenic Drainage Group (Active Comparator): Participants in this group received autogenic drainage as an airway clearance technique for four weeks.
  Interventions: Behavioral: Autogenic Drainage

INTERVENTIONS:
Device: Oscillating Positive Expiratory Pressure Therapy — Oscillating positive expiratory pressure therapy was administered using a handheld device to facilitate airway clearance by providing expiratory resistance and oscillations during exhalation. The intervention was applied for four weeks.
  Arms: Oscillating Positive Expiratory Pressure Therapy Group
Behavioral: Autogenic Drainage — Autogenic drainage is a breathing technique involving controlled breathing at different lung volumes to mobilize and clear bronchial secretions. Participants performed autogenic drainage sessions for four weeks.
  Arms: Autogenic Drainage Group

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a long-term lung condition that causes breathing difficulty, cough, and sputum production. Airway clearance techniques are commonly used to help reduce symptoms and improve breathing in patients with COPD.

This study compared two airway clearance methods-oscillating positive expiratory pressure (OPEP) therapy and autogenic drainage-to determine which method is more effective in improving lung function, sputum clearance, shortness of breath, and quality of life in patients with COPD.

Participants were divided into two groups and received either OPEP therapy or autogenic drainage for four weeks. Outcomes were measured at the beginning of the study and again after completion of the intervention. The findings of this study aim to support evidence-based physiotherapy management for patients with COPD.

DETAILED DESCRIPTION:
This study was a comparative interventional clinical trial conducted to evaluate the effects of oscillating positive expiratory pressure therapy versus autogenic drainage in patients diagnosed with Chronic Obstructive Pulmonary Disease. Ethical approval was obtained from the institutional ethics review committee prior to study initiation, and written informed consent was obtained from all participants.

Eligible participants with stable COPD were enrolled and allocated into two intervention groups. Baseline assessments were performed prior to the initiation of treatment. Participants in the first group received oscillating positive expiratory pressure therapy as part of their airway clearance regimen, while participants in the second group were treated using autogenic drainage techniques. Both interventions were administered over a four-week period.

Outcome measures were assessed at two time points: baseline (pre-intervention) and after completion of the four-week intervention period. Pulmonary function was evaluated using spirometry. Sputum clearance was assessed using the Breathlessness Cough Sputum Scale (BCSS). Dyspnea was measured using the Modified Borg Dyspnea Scale, and quality of life was assessed using the COPD Assessment Test (CAT).

The results of this study aim to compare the effectiveness of the two airway clearance techniques and provide evidence to guide clinical decision-making in the physiotherapy management of patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35 and 50 years
* Both genders
* Participants must have a confirmed diagnosis of Chronic Obstructive Pulmonary Disease (COPD) based on the GOLD 2023 guidelines
* Clinically stable
* History of Sputum Culture

Exclusion Criteria:

* Acute exacerbation of COPD
* Severe cardiovascular, neurological, or musculoskeletal disorders
* Recent thoracic or abdominal surgery
* Presence of other significant respiratory diseases
* Unwillingness to participate or inability to comply with the study protocol

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Change in Forced Expiratory Volume in 1 Second (FEV₁ % Predicted) | Baseline and at 4 weeks
  Pulmonary function was assessed using spirometry by measuring forced expiratory volume in one second (FEV₁), expressed as percentage of the predicted value, in patients with Chronic Obstructive Pulmonary Disease.

SECONDARY OUTCOMES:
Change in Sputum Clearance as Measured by the Breathlessness, Cough, and Sputum Scale (BCSS) | Baseline and at 4 weeks
  Sputum clearance was assessed using the Breathlessness, Cough, and Sputum Scale (BCSS). The BCSS is a patient-reported outcome measure consisting of three items (breathlessness, cough, and sputum), each scored from 0 to 4, resulting in a total score range of 0 to 12. Higher scores indicate worse symptoms.
Change in Dyspnea Severity as Measured by the Modified Borg Dyspnea Scale | Baseline and at 4 weeks
  Dyspnea severity was assessed using the Modified Borg Dyspnea Scale, a numerical rating scale ranging from 0 to 10, where 0 represents no breathlessness and 10 represents maximal breathlessness. Higher scores indicate greater perceived dyspnea.
Change in Health-Related Quality of Life as Measured by the COPD Assessment Test (CAT) | Baseline and at 4 weeks
  Health-related quality of life was assessed using the COPD Assessment Test (CAT), an 8-item questionnaire with total scores ranging from 0 to 40. Higher scores indicate worse health status and greater impact of COPD on daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Hashim, DPT, Principal Investigator — Department of Physical Therapy, The University of Lahore
Locations (1):
- University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because this study was conducted as an academic research project. The informed consent obtained from participants did not include provisions for public data sharing, and the dataset contains sensitive personal health information. Data will be stored securely and used only for academic and research purposes in accordance with institutional ethics approval.

REFERENCES:
- [Background] Bridges, C., Graham-Wollard, L., Morris, H., Annandale, J., & Lewis, K. (2023). S56 A feasibility randomised control trial (RCT) of OPEP verses active cycle of breathing technique (ACBT) in people with chronic obstructive pulmonary disease (COPD). In: BMJ Publishing Group Ltd.
- [Background] Boers, E., Barrett, M., Su, J. G., Benjafield, A. V., Sinha, S., Kaye, L., Zar, H. J., Vuong, V., Tellez, D., Gondalia, R., Rice, M. B., Nunez, C. M., Wedzicha, J. A., & Malhotra, A. (2023). Global Burden of Chronic Obstructive Pulmonary Disease Through 2050. JAMA Netw Open, 6(12), e2346598. https://doi.org/10.1001/jamanetworkopen.2023.46598
- [Background] Bishop, K. L., & Malone, D. J. (2024). Pulmonary Diseases and Disorders. In Acute Care Physical Therapy (pp. 245-310). Routledge.
- [Background] Belli, S., Prince, I., Savio, G., Paracchini, E., Cattaneo, D., Bianchi, M., Masocco, F., Bellanti, M. T., & Balbi, B. (2021). Airway clearance techniques: the right choice for the right patient. Frontiers in medicine, 8, 544826.
- [Background] Awokola, B., Amusa, G., Jewell, C., Okello, G., Stobrink, M., Finney, L., Mohammed, N., Erhart, A., & Mortimer, K. (2022). Chronic obstructive pulmonary disease in sub-Saharan Africa. The International Journal of Tuberculosis and Lung Disease, 26(3), 232-242.
- [Background] Alruwaili, A. T. S., Alsirhani, A. F., khlaif Alrwili, A., Aldaghmi, M. T. A., Alharbi, S. E. M., & Aldhafeeri, R. Z. (2024). NURSING, PHYSICAL THERAPY, AND RESPIRATORY CARE IN ENHANCING PHYSICAL AND PSYCHOLOGICAL REHABILITATION FOR PATIENTS WITH RESPIRATORY DISEASES. Gland Surgery, 9(2).
- [Background] Alghamdi, S. M., Alsulayyim, A. S., Alasmari, A. M., Philip, K. E., Buttery, S. C., Banya, W. A., Polkey, M. I., Birring, S. S., & Hopkinson, N. S. (2023). Oscillatory positive expiratory pressure therapy in COPD (O-COPD): a randomised controlled trial. Thorax, 78(2), 136-143.
- [Background] Adeloye, D., Song, P., Zhu, Y., Campbell, H., Sheikh, A., & Rudan, I. (2022). Global, regional, and national prevalence of, and risk factors for, chronic obstructive pulmonary disease (COPD) in 2019: a systematic review and modelling analysis. The Lancet Respiratory Medicine, 10(5), 447-458.